CLINICAL TRIAL: NCT00788125
Title: Dasatinib With Ifosfamide, Carboplatin, Etoposide: A Pediatric Phase I/II Trial
Brief Title: Dasatinib, Ifosfamide, Carboplatin, and Etoposide in Treating Young Patients With Metastatic or Recurrent Malignant Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated early due a shift in resources after lackluster performance of the drug.
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 07053; P30CA033572 (NIH); CHNMC-07053; CA180 121; CDR0000617760 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Results first posted 2022-04-27 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Brain and Central Nervous System Tumors; Childhood Germ Cell Tumor; Extragonadal Germ Cell Tumor; Kidney Cancer; Liver Cancer; Lymphoma; Neuroblastoma; Ovarian Cancer; Sarcoma; Testicular Germ Cell Tumor; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: previously treated childhood rhabdomyosarcoma; metastatic childhood soft tissue sarcoma; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; metastatic osteosarcoma; recurrent childhood rhabdomyosarcoma; recurrent childhood soft tissue sarcoma; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent osteosarcoma; unspecified childhood solid tumor, protocol specific; recurrent Wilms tumor and other childhood kidney tumors; recurrent neuroblastoma; stage 4S neuroblastoma; childhood extracranial germ cell tumor; childhood malignant ovarian germ cell tumor; childhood malignant testicular germ cell tumor; childhood teratoma; clear cell sarcoma of the kidney; childhood renal cell carcinoma; recurrent renal cell cancer; congenital mesoblastic nephroma; cystic nephroma; peripheral primitive neuroectodermal tumor of the kidney; rhabdoid tumor of the kidney; disseminated neuroblastoma; recurrent malignant testicular germ cell tumor; recurrent ovarian germ cell tumor; recurrent childhood liver cancer; stage IV childhood liver cancer; angioimmunoblastic T-cell lymphoma; stage IV childhood Hodgkin lymphoma; stage IV childhood large cell lymphoma; stage IV childhood lymphoblastic lymphoma; stage IV childhood small noncleaved cell lymphoma; recurrent childhood grade III lymphomatoid granulomatosis; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent/refractory childhood Hodgkin lymphoma; childhood diffuse large cell lymphoma; childhood grade III lymphomatoid granulomatosis; childhood immunoblastic large cell lymphoma; childhood nasal type extranodal NK/T-cell lymphoma; Burkitt lymphoma; recurrent childhood anaplastic large cell lymphoma; stage IV childhood anaplastic large cell lymphoma; childhood central nervous system choriocarcinoma; childhood central nervous system embryonal tumor; childhood central nervous system germ cell tumor; childhood central nervous system germinoma; childhood central nervous system mixed germ cell tumor; childhood central nervous system teratoma; childhood central nervous system yolk sac tumor; recurrent childhood central nervous system embryonal tumor; childhood choroid plexus tumor; childhood craniopharyngioma; childhood ependymoblastoma; childhood medulloepithelioma; childhood infratentorial ependymoma; childhood supratentorial ependymoma; childhood oligodendroglioma; childhood pineal parenchymal tumor; childhood grade I meningioma; childhood grade II meningioma; childhood grade III meningioma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood ependymoma; recurrent childhood medulloblastoma; recurrent childhood pineoblastoma; recurrent childhood supratentorial primitive neuroectodermal tumor; recurrent childhood visual pathway and hypothalamic glioma; recurrent uterine sarcoma; childhood high-grade cerebellar astrocytoma; childhood high-grade cerebral astrocytoma; childhood low-grade cerebellar astrocytoma; childhood low-grade cerebral astrocytoma; childhood atypical teratoid/rhabdoid tumor; primary central nervous system non-Hodgkin lymphoma; primary central nervous system Hodgkin lymphoma; childhood extragonadal germ cell tumor; recurrent childhood malignant germ cell tumor; recurrent childhood brain stem glioma; recurrent childhood subependymal giant cell astrocytoma; recurrent childhood brain tumor; recurrent childhood spinal cord neoplasm
MeSH Terms: conditions — Central Nervous System Neoplasms; Kidney Neoplasms; Liver Neoplasms; Lymphoma; Neuroblastoma; Ovarian Neoplasms; Sarcoma; Testicular Germ Cell Tumor; Neuroectodermal Tumors, Primitive, Peripheral; Osteosarcoma; Wilms Tumor; Ovarian Germ Cell Cancer; Testicular Neoplasms; Teratoma; Carcinoma, Renal Cell; Nephroma, Mesoblastic; Immunoblastic Lymphadenopathy; Dendritic Cell Sarcoma, Interdigitating; Burkitt Lymphoma; Recurrence; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Choroid Plexus Neoplasms; Oligodendroglioma; Astrocytoma; Familial ependymoma; Medulloblastoma; Optic Nerve Glioma; Rhabdoid Tumor; Spinal Cord Neoplasms | interventions — Carboplatin; Dasatinib; etoposide phosphate; Ifosfamide; Microarray Analysis; Blotting, Western; Immunohistochemistry; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Level -1: 25 mg/m^2/dose BID PO Dasatinib x 17 days. Period 1: 35 mg/m^2/dose BID PO Dasatinib x 17 days. Period 2: 50 mg/m^2/dose BID PO Dasatinib x 17 days. Period 3: 65 mg/m^2/dose BID PO Dasatinib x 17 days. Period 4: 85 mg/m^2/dose BID PO Dasatinib x 17 days. Period 5 (Dasatinib alone phase only): 110 mg/m^2/dose BID PO. Sponsor withdrew support before a second level could be attempted.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dasatinib with Ifosfamide, Carboplatin, Etoposide (Experimental)
  Interventions: Drug: carboplatin; Drug: dasatinib; Drug: etoposide phosphate; Drug: ifosfamide; Genetic: microarray analysis; Genetic: western blotting; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Procedure: therapeutic conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Drug: carboplatin
Drug: dasatinib
Drug: etoposide phosphate
Drug: ifosfamide
Genetic: microarray analysis
Genetic: western blotting
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: therapeutic conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs in chemotherapy, such as ifosfamide, carboplatin, and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving dasatinib together with ifosfamide, carboplatin, and etoposide may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of dasatinib when given together with ifosfamide, carboplatin, and etoposide and to see how well they work in treating young patients with metastatic or recurrent malignant solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose (MTD) of dasatinib when given immediately following ifosfamide, carboplatin, and etoposide phosphate (D-ICE) as a re-induction regimen in young patients with metastatic or recurrent malignant solid tumors. (Phase I)
* To describe and define the toxicities of D-ICE in these patients. (Phase I)
* To determine the safety and feasibility of prolonged administration of single-agent dasatinib following completion of 2-6 courses of D-ICE in these patients. (Phase I)
* To estimate the overall survival, progression-free survival, and time to progression in patients treated with D-ICE at the MTD followed by single-agent dasatinib. (Phase II)
* To estimate the response rate to two courses of D-ICE when given at the MTD in these patients. (Phase II)

Secondary

* To determine the phosphotyrosine state of SRC family kinases and related signaling pathways, including FAK, STAT3, VEGFR, AKT, EGFR, KIT, EPHA2, and PDGFR, in paraffin-embedded tumor samples as measured by immunohistochemistry prior to and during treatment with dasatinib.
* To assess gene expression profiling in fresh frozen tissue samples as measured by microarray analysis (Affymetrix GeneChips) at baseline to identify molecular signatures that may predict response to dasatinib.
* To correlate biomarkers and molecular signatures with dasatinib dosage, toxicity, and antitumor activity.
* To evaluate the effect of dasatinib on phosphorylation of SRC family kinases in peripheral blood mononuclear cell samples as a surrogate marker of response prior to treatment with dasatinib, at days 14-21 or when WBC ≥ 500/μL, during each treatment course, at the time of local control, and at the time of progression.

OUTLINE: This is a multicenter, phase I, dose-escalation study of dasatinib followed by a phase II study. Patients enrolled in phase II are stratified according to disease.

Patients receive D-ICE comprising oral dasatinib twice daily on days 5-21, ifosfamide IV over 1 hour and etoposide phosphate IV over 1 hour on days 1-5, and carboplatin IV over 1 hour on days 1 and 2. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo radiotherapy and/or surgery (consolidation therapy) after 2, 4, or 6 courses of D-ICE. After completion of consolidation therapy, patients receive oral dasatinib twice daily for up to 6 months in the absence of disease progression or unacceptable toxicity.

Tumor tissue and peripheral blood mononuclear cell (PBMC) samples are collected periodically for correlative laboratory studies. PBMCs are analyzed by western blotting for total and phospho-SRC, phospho-FAK, and other relevant biomarkers. Tumor tissue samples are analyzed by IHC for total and phospho-SRC, phospho-FAK, phospho-STAT3, phospho-KIT, and phospho-PDGFR, EPHA2, and VEGF. Tumor tissue samples are also analyzed by microarray gene expression profiling to define a potential molecular signature or gene expression pattern that may predict response to dasatinib.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant solid tumor that did not respond to or relapsed after standard first-line chemotherapy or other antineoplastic therapy (if the standard therapy for the tumor is generally recognized to be beneficial)

  * Must have been initially diagnosed with malignancy prior to 25 years of age
  * Radiographic, nuclear image, or biopsy confirmation of disease within the past 4 weeks
* Meets one of the following criteria:

  * Phase I: Relapsed/refractory malignant solid tumor (excluding CNS tumors)

    * Patients with recurrent or metastatic disease that was completely resected just prior to study entry are eligible
  * Phase II: Patients are stratified according to one of the following diagnoses:

    * Stratum A: Relapsed sarcoma (rhabdomyosarcoma, osteosarcoma, or Ewing sarcoma)
    * Stratum B: Other relapsed solid tumors, including any of the following:

      * Other soft tissue sarcomas
      * Kidney tumors
      * Lymphoma
      * CNS tumors*
      * Other solid tumors (neuroblastoma, gonadal and germ cell tumors, liver tumors, or miscellaneous tumors)
    * Stratum C: Newly diagnosed, poor-risk metastatic sarcoma consisting of unresectable pulmonary metastases (≥ 6 nodules) and/or disease involving multiple bones or other organs NOTE: *Patients with recurrent primary CNS tumors are eligible for the phase II portion of this study provided there are no significant intratumoral bleeding toxicities seen in either COG pediatric phase I studies of dasatinib or the phase I portion of this study
* Radiographically measurable disease (Phase II)

  * Measurable disease is not required for patients who are enrolled in the phase I portion of this study
* No bone marrow involvement (Phase I)

  * Patients with bone marrow involvement are eligible for the phase II portion of this study provided they are not known to be refractory to red cell or platelet transfusions

PATIENT CHARACTERISTICS:

* Lansky performance status (PS) 50-100% (patients 1-16 years of age) or Karnofsky PS 50-100% (patients > 16 years of age)
* Life expectancy ≥ 8 weeks
* ANC > 1,000/μL
* Platelet count > 75,000/μL
* Creatinine clearance or GFR ≥ 70 mL/min OR creatinine < 1.5 times upper limit of normal (ULN)
* Bilirubin < 1.5 times ULN for age
* SGOT or SGPT < 2.5 times ULN for age (< 5 times ULN if liver involvement by tumor)
* Ejection fraction normal by MUGA OR shortening fraction > 28%
* No evidence of cardiac arrhythmias requiring therapy
* Corrected QTc interval < 450 msecs
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to comply with the safety monitoring requirements of this study
* No uncontrolled infection
* No swallowing dysfunction that would preclude oral medication intake

  * Gastric or jejunal tube allowed provided it is functioning
* No history of significant bleeding disorder unrelated to cancer, including the following:

  * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
  * Acquired bleeding disorder diagnosed within the past year (e.g., acquired anti-factor VIII antibodies)
  * Ongoing or recent (within the past 3 months) significant gastrointestinal bleeding

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior therapy
* At least 7 days since prior and no concurrent drugs known to cause Torsades de Pointes, including the following:

  * Procainamide or disopyramide
  * Amiodarone, sotalol, ibutilide, or dofetilide
  * Erythromycin or clarithromycin
  * Chlorpromazine, haloperidol, mesoridazine, or thioridazine
  * Bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, or lidoflazine
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosourea-containing therapy)
* At least 3 months since prior ifosfamide, carboplatin, and/or etoposide phosphate in the exact combination and dosage as administered in this study
* More than 7 days since prior filgrastim (G-CSF), sargramostim (GM-CSF), or interleukin-11
* More than 14 days since prior pegfilgrastim
* More than 30 days since prior epoetin alfa
* No prior cranial-spinal irradiation at doses > 2,400 cGy
* No prior radiotherapy, including total-body irradiation, to > 50% of the bone marrow space
* No other concurrent investigational drugs or anticancer agents
* No concurrent enzyme-inducing anticonvulsants (e.g., phenytoin, phenobarbital, felbamate, primdone, oxcarbazepine, or carbamazepine)
* No concurrent anti-thrombotic or anti-platelet agents (e.g., warfarin, heparin, low molecular weight heparin, aspirin, ibuprofen, or other NSAIDs)
* No concurrent CYP3A4 inhibitors (e.g., itraconazole, ketoconazole, or voriconazole)
* No concurrent highly active antiretroviral therapy for HIV-positive patients
* No concurrent St. John's wort
* No IV bisphosphonates during the first 8 weeks of dasatinib therapy

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2008-09-03 (Actual); Primary Completion 2010-04-30 (Actual); Study Completion 2022-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith K. Sato, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://clinicaltrials.gov/ct2/show/NCT00788125

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase I study participants were recruited based on physician referral at City of Hope Medical Center, between September 04, 2008 and February 04, 2010. Seven patients met the inclusion criteria and were enrolled on the study.
Pre-assignment Details: Phase I of this study involved City of Hope patients, only. This protocol did not progress beyond Period 1: 35 mg/m^2/dose BID to other dose levels within Phase I. This protocol did not progress to Phase II, which would have involved other institutions. Sponsor withdrew support.
Groups:
- Period 1: 35 mg/m^2 Dasatinib BID PO: 35 mg/m^2/dose BID PO Dasatinib x 17 days
  Ifosfamide, Carboplatin, Etoposide
  microarray analysis
  western blotting
  immunohistochemistry staining method
  laboratory biomarker analysis
  therapeutic conventional surgery
  radiation therapy
Period: Overall Study
Arm/Group | Period 1: 35 mg/m^2 Dasatinib BID PO
Started | 7
Completed | 1
Not Completed | 6
Not completed — Death | 6

BASELINE CHARACTERISTICS:
Groups:
- Period 1: 35 mg/m^2 Dasatinib BID PO: 35mg/m^2/dose BID PO Dasatinib x 17 days
  Ifosfamide, Carboplatin, Etoposide
  microarray analysis
  western blotting
  immunohistochemistry staining method
  laboratory biomarker analysis
  therapeutic conventional surgery
  radiation therapy
Arm/Group | Period 1: 35 mg/m^2 Dasatinib BID PO
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 14.6 [4.8 to 26.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Maximum Administered Dose of Dasatinib (Phase I)
Description: This field captured the maximum dose of dasatinib administered.
Time Frame: 28 days after start of course 1
Population: Level -1: 25 mg/m^2/dose BID PO Dasatinib x 17 days. Period 1: 35 mg/m^2/dose BID PO Dasatinib x 17 days. Period 2: 50 mg/m^2/dose BID PO Dasatinib x 17 days. Period 3: 65 mg/m^2/dose BID PO Dasatinib x 17 days. Period 4: 85 mg/m^2/dose BID PO Dasatinib x 17 days. Period 5 (Dasatinib alone phase only): 110 mg/m^2/dose BID PO. Sponsor withdrew support before a second level could be attempted.
Measure: Number; unit: mg/m2 dose BID
Groups:
- Period 1: 35 mg/m^2/Dose BID PO Dasatinib x 17 Days: 35 mg/m^2/dose BID PO Dasatinib x 17 days
  Ifosfamide, Carboplatin, Etoposide
  therapeutic conventional surgery
  radiation therapy
Arm/Group | Period 1: 35 mg/m^2/Dose BID PO Dasatinib x 17 Days
Number analyzed (Participants) | 7
mg/m2 dose BID | 35

ADVERSE EVENTS:
Time Frame: Adverse events were collected for twenty-eight days post-first administration of Dasatinib, plus 14 days, to equal 42 days of follow-up for toxicity. After two months of follow-up of a three-patient cohort, consideration would be made for escalating the dose level in the next cohort of three patients. If toxicity does not resolve to meet study parameters for re-treatment by day 42 of the course, the patient must be removed from the study.
Groups:
- Period 1: 35 mg/m^2 Dasatinib BID PO: 35mg/m^2/dose BID PO Dasatinib x 17 days
  Iphosfamide, Carboplatin, Etoposide
  microarray analysis
  western blotting
  immunohistochemistry staining method
  laboratory biomarker analysis
  therapeutic conventional surgery
  radiation therapy
Arm/Group | Period 1: 35 mg/m^2 Dasatinib BID PO
All-Cause Mortality (participants affected / at risk) | 6/7
Serious Adverse Events (participants affected / at risk) | 6/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: 35 mg/m^2 Dasatinib BID PO (N=7)
Infection -- Brain (encephalitis, infections) (Infections and infestations) | 1 — Grade 5 Infection (documented clinically or microbiologically) with grade 3 or 4 neutrophils(ANC<1.0 x 10e9/L) -- Brain (encephalitis, infections) Possibly, probably, or definitely attributable to the study regimen.
Death not associated with CTCAE term -- Death NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 — Attribution is: Unlikely or unrelated to the study regimen.
Death not associated with CTCAE term -- Disease progression, NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 — Attributed is: Unlikely or unrelated to the study regimen.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: 35 mg/m^2 Dasatinib BID PO (N=7)
Allergic reaction/hypersnsitivity (including drug fever) (Immune system disorders) | 2
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 6
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 6
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 6
Platelets (Blood and lymphatic system disorders) | 6
Palpitations (Cardiac disorders) | 1
Supraventricular and nodal arrhythmia (Cardiac disorders) | 5
Vasovagal episode (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 4
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Pericardial effusion (non-malignant) (Cardiac disorders) | 1
INR (International Normalized Ratio of prothrombin time) (Vascular disorders) | 1
PTT (Partial Thromboplastin Time) (Vascular disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 5
Fever (absent of neutropenia, ANC<1.0E9/L) (General disorders) | 4
Insomnia (General disorders) | 1
Rigors/chills (General disorders) | 4
Sweating (diaphoresis) (General disorders) | 1
Weight gain (General disorders) | 2
Weight loss (General disorders) | 2
Bruising (in abscence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 3
Acne (Skin and subcutaneous tissue disorders) | 1
Blue Skin (Skin and subcutaneous tissue disorders) | 1
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 1
Discoloration (Skin and subcutaneous tissue disorders) | 1
Pale (Skin and subcutaneous tissue disorders) | 1
Blue (Skin and subcutaneous tissue disorders) | 1
Skin Irritation (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 4
Flushing (Skin and subcutaneous tissue disorders) | 1
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 5
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 5
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4
Cushingoid appearance (e.g. moon face, buffalo hump, centripetal obesity, cutaneous striae) (Endocrine disorders) | 1
Anorexia (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 5
Distension/bloating, abdominal (Gastrointestinal disorders) | 2
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 2
Esophagitis (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 3
Heartburn/dyspepsia (Gastrointestinal disorders) | 1
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 4
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 6
Salivary gland changes/saliva (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Hematoma (Vascular disorders) | 3
Hemorrhage, GI (Vascular disorders) | 2
Hemorrhage, GU (Vascular disorders) | 2
Hemorrhage, pulmonary/upper respiratory (Vascular disorders) | 3
Hemorrhage/Bleeding -- Other, Conjunctival (Vascular disorders) | 1
Hemorrhage/Bleeding -- Other, Scleral (Vascular disorders) | 1
Febrile neutropenia ANC<1E9/L (fever of unknown origin without documented infection) (Infections and infestations) | 2
Infection with Gr 3 or 4 neutrophils (ANC<1E9/L) (Infections and infestations) | 5
Infection with normal ANC or Grade 1 or 2 neutrophil (Infections and infestations) | 1
Edema: head and neck (Blood and lymphatic system disorders) | 2
Edema: limb (Blood and lymphatic system disorders) | 3
Edema: trunk/genital (Blood and lymphatic system disorders) | 3
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 5
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 5
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 6
Alkaline phosphatase (Metabolism and nutrition disorders) | 3
Alkalosis metabolic or respiratory) (Metabolism and nutrition disorders) | 1
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 6
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 5
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 1
Creatinine (Metabolism and nutrition disorders) | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 2
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 5
Metabolic/Laboratory -- Other: Hematochromatomatosis (Metabolism and nutrition disorders) | 1
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 6
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 6
Proteinuria (Metabolism and nutrition disorders) | 3
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 6
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 5
Muscle weakness, not due to neuropathy, Extremity Lower (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness, not due to neuropathy, Extremity Upper (Musculoskeletal and connective tissue disorders) | 1
Muscular/skeletal hypoplasia (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/Soft Tissue, Other: Atrophy (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/Soft Tissue, Other: Avulsion (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/Soft Tissue, Other: Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Ataxia (incoordination) (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 3
Memory Impairment (Nervous system disorders) | 2
Mood alteration (Psychiatric disorders) | 5
Mood alteration, depression (Psychiatric disorders) | 1
Personality/behavioral (Psychiatric disorders) | 1
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 1
Somnolescence/depressed level of consciousness (Nervous system disorders) | 3
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1
Syncope (fainting) (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Dry eye syndrome (Eye disorders) | 1
Ocular/visual, other: Conjunctivitis (Eye disorders) | 1
Pain (General disorders) | 6
Pain, other: Cathetar related (General disorders) | 1
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory, Other: Phrenic Nerve Cut (Respiratory, thoracic and mediastinal disorders) | 1
Bladder spasms (Renal and urinary disorders) | 1
Incontinence, urinary (Renal and urinary disorders) | 2
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1
Urine color change (Renal and urinary disorders) | 1
Petechiae/purpura (hemorrhage/bleeding into the skin or mucosa) (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2009-12-08): https://cdn.clinicaltrials.gov/large-docs/25/NCT00788125/Prot_SAP_000.pdf